CLINICAL TRIAL: NCT04739072
Title: Minimal Residual Disease Assessment in Colorectal Cancer (MiRDA-C)
Brief Title: Minimal Residual Disease Assessment in Patients With Colorectal Cancer, the MiRDA-C Study
Status: Recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: PA18-1171; NCI-2020-10034 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); PA18-1171 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2021-02-02; First posted 2021-02-04 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-11

CONDITIONS: Colorectal Adenocarcinoma; Stage I Colorectal Cancer AJCC v8; Stage II Colorectal Cancer AJCC v8; Stage IIA Colorectal Cancer AJCC v8; Stage IIB Colorectal Cancer AJCC v8; Stage IIC Colorectal Cancer AJCC v8; Stage III Colorectal Cancer AJCC v8; Stage IIIA Colorectal Cancer AJCC v8; Stage IIIB Colorectal Cancer AJCC v8; Stage IIIC Colorectal Cancer AJCC v8; Stage IV Colorectal Cancer AJCC v6; Stage IVA Colorectal Cancer AJCC v8; Stage IVB Colorectal Cancer AJCC v8; Stage IVC Colorectal Cancer AJCC v8
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ancillary-correlative (biospecimen collection): Patients undergo collection of blood samples at baseline, during each neoadjuvant therapy treatment, prior to surgical resection, and up to 4 times per year for up to 5 years. Patients also undergo collection of tissue sample at time of surgical resection. Patients medical records may also be reviewed.
  Interventions: Procedure: Biospecimen Collection; Other: Electronic Health Record Review

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of blood and tissue samples
Other: Electronic Health Record Review — Review of medical records

SUMMARY:
This study investigates if circulating tumor DNA (ctDNA) and other tumor-related molecules/chemicals released in the blood can help doctors predict if colorectal cancer may come back or spread. Tumors shed DNA and other cancer related chemicals into the blood that can be identified and studied further to provide information about the cancer. Information gathered from this study may help researchers better understand if ctDNA found in the blood can predict whether colorectal cancer may come back or spread.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Demonstrate ability to monitor cancer-specific deoxyribonucleic acid (DNA), ribonucleic acid (RNA), and proteomic alterations from plasma.

II. Improve detection of recurrences post completion of curative therapies through monitoring of plasma cancer-specific DNA, RNA and proteomic alterations.

SECONDARY OBJECTIVES:

I. Qualitative and quantitative changes in cancer-specific plasma alterations during neoadjuvant, adjuvant therapies and surveillance.

II. Disease free survival (DFS) of patients with detectable cancer-specific plasma alterations.

III. Overall survival (OS) of patients with detectable cancer-specific plasma alterations.

EXPLORATORY OBJECTIVES:

I. Optimal combination of cancer-specific plasma DNA, RNA and / or proteomic alterations for early detection of recurrences.

II. Sensitivity, specificity, positive predictive and negative predictive values of cancer-specific plasma alterations in detecting recurrences.

III. Correlation between cancer-specific alterations in plasma and tissue and either with outcomes including DFS & OS.

IV. Nature and frequency of detection of incidental non-colorectal cancer related DNA, RNA and / or proteomic alterations.

OUTLINE:

Patients undergo collection of blood samples at baseline, during each neoadjuvant therapy treatment, prior to surgical resection, and up to 4 times per year for up to 5 years. Patients also undergo collection of tissue sample at time of surgical resection. Patients' medical records may also be reviewed.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. Histological/cytological confirmation of colorectal adenocarcinoma.
3. Patients with any stage colorectal adenocarcinoma deemed potentially eligible for curative intent treatment. Patients with stages II-IV colorectal cancer post-R0 resection may also be enrolled onto the protocol any time before or up to 3 months post-surgery and prior to initiating adjuvant therapy.
4. Ability to understand and the willingness to sign a written informed consent document.
5. Willing to pursue standard of care surveillance post completion of curative therapies.
6. Willing to provide blood samples for correlative research.

Exclusion Criteria:

1. Known active malignancies other than colorectal adenocarcinoma that may interfere with detection and / or interpretation of circulating plasma markers. Patients with known clonal hematopoiesis of indeterminate potential are eligible.
2. Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with colorectal cancer at MD Anderson Cancer Center.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2019-11-22 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Analysis of deoxyribonucleic (DNA), ribonucleic acid (RNA), and proteomic alterations from plasma | Up to 5 years
  To detect circulating tumor DNA (ctDNA) in plasma samples from patients with colorectal cancer (CRC) who have completed curative therapies (i.e. minimal residual disease) towards predicting recurrence earlier than the current standard of care utilizing the CRC23 assay and the LUNAR assay from Guardant Health technology.
Detection of recurrences post completion of curative therapies | Up to 5 years
  To detect ctDNA in plasma samples from patients with CRC who have completed curative therapies (i.e. minimal residual disease) towards predicting recurrence earlier than the current standard of care utilizing the CRC23 assay and the LUNAR assay from Guardant Health technology.

SECONDARY OUTCOMES:
Changes in cancer-specific plasma alterations during neoadjuvant, adjuvant therapies and surveillance | Baseline up to 5 years
  Will assess the association between changes in circulating molecules and response in patients undergoing neoadjuvant therapy by linear or logistic regression models
Disease free survival (DFS) | Up to 5 years
Overall survival (OS) | Up to 5 years

OTHER OUTCOMES:
Optimal combination of cancer-specific plasma DNA, RNA and / or proteomic alterations for early detection of recurrences | Up to 5 years
Sensitivity, specificity, positive predictive and negative predictive values of cancer-specific plasma alterations in detecting recurrences | Up to 5 years
Correlation between cancer-specific alterations in plasma and tissue and either with outcomes including DFS & OS | Up to 5 years
Nature and frequency of detection of incidental non-colorectal cancer related DNA, RNA and / or proteomic alterations | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Arvind Dasari, Principal Investigator — M.D. Anderson Cancer Center
Locations (10):
- United States (10):
  - Banner - MD Anderson Cancer Center, Gilbert, Arizona
  - Baptist- MD Anderson Cancer Center, Jacksonville, Florida
  - The Queen's Medical Center, Honolulu, Hawaii
  - St. Luke's Cancer Institute, Boise, Idaho
  - Cooper Hospital UNIV MED CTR., Camden, New Jersey
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Houston Methodist Cancer Center, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - UT Health San Antonio MD Anderson Cancer Center, San Antonio, Texas
  - Baylor Scott & White Research Institute, Temple, Texas

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org